CLINICAL TRIAL: NCT03672383
Title: Randomized, Controlled, Observer-blinded, Intra-individual Clinical Trial to Examine the Efficacy and Safety of a New Medical Device (Modified Diprobase Formulation) in Adults With Quiescent Atopic Dermatitis
Brief Title: Functional Study to Investigate the Efficacy of a New Medical Device (Modified Diprobase Formulation)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19689
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Observer-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY987534 (Treated Arm) (Experimental): Subjects with quiescent atopic dermatitis. Right or left volar forearm with test product applied.
  Interventions: Device: BAY987534
- Untreated Arm (No Intervention): Subjects with quiescent atopic dermatitis. Right or left volar forearm without test product applied.

INTERVENTIONS:
Device: BAY987534 — Form: cream; Route of Administration: topical; Frequency of Administration: twice daily ; Duration of Treatment: 4 weeks .
  Other Names: modified Diprobase formulation
  Arms: BAY987534 (Treated Arm)

SUMMARY:
This clinical trial is intended to investigate the efficacy and safety of a medical device compared to untreated on patients with quiescent atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients being willing and able to provide written informed consent to participate in the study;
* Patients with self-reported history of AD (at least one flare up in the past with mild to moderate intensity), but with no flare-up within the last month;
* Patients aged between 18 - 65 years;
* Corneometer value < 35 a.u (on one volar forearm);
* Skin type I-IV (Fitzpatrick et al. 1974);
* Patients willing to adhere to trial procedures;
* Patients willing to discontinue the use of own cleansing and cosmetic products (e.g. soaps, creams, moisturizers) in test areas 3 days before Day 1 and throughout the course of the trial;
* Patients willing to stop smoking 2 hours before the instrumental measurements;
* Patients willing not to drink caffeinated beverages 2 hours before the instrumental measurements;
* Patients willing to avoid contact with water in the test areas 2 hours before the instrumental measurements;
* Negative urine pregnancy test (for female patients of child bearing potential);
* Women of child bearing potential have to use reliable methods of contraception with a low failure rate (i.e., less than 1 % per year; implants, injectables, combined oral contraceptives, hormone-based intrauterine-devices, sexual abstinence or vasectomized partner).

Exclusion Criteria:

* Any other skin disease on the whole body that would interfere the clinical assessment in the opinion of the Investigator;
* Intake of drugs interfering with the immune system (e.g. corticosteroids, immunosuppressive drugs and antihistamines) within 30 days before screening as well as during the trial (with exception of routine vaccinations);
* Intrarectal or topical corticosteroids (in the test area) within 2 weeks before screening as well as during the trial;
* Known allergies to any of the ingredients of the test product;
* Any use of another topical emollient or other established treatment for atopic dermatitis in the test area;
* Any other adjuvant therapy for atopic dermatitis (UV therapy, probiotics homeopathy etc.);
* Patients with a Body Mass Index > 30;
* Diabetes mellitus;
* Patients who use tanning beds regularly within the past 2 years;
* Exposure of the test area to the sun;
* Pregnant or lactating women;
* Moles, tattoos, pigmentation or scars on the forearms that would influence the instrumental measurements;
* Hairy skin on test areas;
* Patients with psychiatric conditions that might limit the participation in the trial and/or that lead to the assumption that the ability to completely understand the consequences of consent is missing;
* Patients with any history of drug addiction or alcoholism in the past 3 years;
* Patients with expected poor compliance;
* Patients, who are inmates of psychiatric wards, prison or state institutions;
* Participation in a clinical trial with investigational medicinal products or medical devices within the last 30 days prior to the start of this trial;
* Patients underlying any other restrictions due to the participation in other tests / at other test institutes;
* Employees of the trial sites or of the Sponsor's company;
* Patients that according to the opinion of the Investigator should not participate in the trial for any reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
AUC of the skin hydration assessed of treatment with the test product compared to untreated | Up to 4 weeks
  AUC: Area under the curve

SECONDARY OUTCOMES:
AUC of the short term skin hydration | Day 1
  Comparison of the test product to untreated
Skin hydration by measuring skin capacitance assessed by Corneometry (unit: a.u.) | Up to 4 weeks
  Comparison of the test product to untreated based on differences to Baseline as well as the comparison to Baseline
Skin hydration after treatment by measuring skin capacitance assessed by Corneometry (unit: a.u.) | Up to 4 weeks
  a.u.: arbitrary units
Skin pH | Up to 4 weeks
  Comparison of the test product to untreated based on the differences to Baseline
Transepidermal water loss | Up to 4 weeks
  Comparison of the test product to untreated based on differences to Baseline for SDS (Sodium dodecyl sulfate) unchallenged and SDS challenged skin
Stratum corneum thickness assessed by Raman Spectrometry (unit: µm) | Up to 8 hours
  Comparison of the test product to untreated
Water gradient within stratum corneum assessed by Raman Spectrometry | Up to 8 hours
  Comparison of the test product to untreated
Number of participants with adverse events (AEs) | Up to 4 weeks
Compliance check | Day 29
  The diaries will be collected and checked for compliance and completeness of the daily record
Water content within stratum corneum assessed by Raman Spectrometry (unit: %) | Up to 8 hours
  Comparison of the test product to untreated

CONTACTS AND LOCATIONS:
Locations (1):
- proDerm, Hamburg, Germany

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/